CLINICAL TRIAL: NCT05112094
Title: Therapeutic Effect of Peripheral Magnetic Stimulation Generated by the Super-inductive System to Treat Patient With Post-stroke Shoulder-hand Syndrome
Brief Title: Peripheral Magnetic Stimulation to Treat Patient With Post-stroke Shoulder-hand Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202105016RIPB
Record Dates: First submitted 2021-10-03; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-07

CONDITIONS: Reflex Sympathetic Dystrophy of Upper Limb; Stroke
Keywords: shoulder pain; magnetic stimulation; electric stimulation; reflex sympathetic dystrophy
MeSH Terms: conditions — Reflex Sympathetic Dystrophy; Stroke; Shoulder Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- peripheral magnetic stimulation (Experimental): peripheral magnetic stimulation (50-80% output, 20-40Hz, pulse duration 3-5 seconds, for 15 minutes) + physical therapy (shoulder range of motion exercise and stretching 30-40 minutes per day)
  Interventions: Device: peripheral magnetic stimulation; Other: physical therapy
- physical therapy only (Placebo Comparator): regular physical therapy (shoulder range of motion exercise and stretching 30-40 minutes per day)
  Interventions: Other: physical therapy

INTERVENTIONS:
Device: peripheral magnetic stimulation — peripheral magnetic stimulation at ipsilateral shoulder ((50-80% output, 20-40Hz, pulse duration 3-5 seconds, for 15 minutes) ) + regular physical therapy(shoulder range of motion exercise and stretching 30-40 minutes per day)
  Arms: peripheral magnetic stimulation
Other: physical therapy — regular physical therapy(shoulder range of motion exercise and stretching 30-40 minutes per day)

SUMMARY:
Shoulder-hand syndrome is a common complication following stroke, constituting of excessive pain, swelling, heat, limited range of motion, and trophic change of the affected limbs. It not only has an extensive negative impact on both physical and psychological aspects of a stroke patient's well-being, but also impose burden on the health care system and the patient's family. Despite its relatively high incidence, there is neither well-established treatment protocol, nor high quality evidence for a single effective treatment. The objective of the present study is to investigate the efficacy, including pain, spasticity, and subluxation reduction, muscle strengthening, and shoulder range of motion improvement, of high-intensity peripheral magnetic stimulation generated by the super-inductive system to treat patients with post-stroke shoulder-hand syndrome.

DETAILED DESCRIPTION:
The present study aims to investigate the therapeutic effects achieved by the peripheral magnetic stimulation for treating post-stroke shoulder-hand syndrome. The investigators plan to use high-intensity peripheral magnetic stimulation generated by the super-inductive system for treatment of post-stroke shoulder-hand syndrome. In terms of study design, the treatment group will receive 10 sessions of high-intensity peripheral magnetic stimulation 5 days a week for 2 weeks, with physical and occupational therapy kept as usual; while the control group will only receive conventional physical and occupational therapy. Comprehensive assessment, including history taking and physical examination testing for muscle strength, spasticity, shoulder range of motion, before and after the intervention will be conducted for evaluation.

ELIGIBILITY:
Inclusion criteria:

* >=20 years old
* Stroke in recent 6 months
* Clear consciousness
* Clinical diagnosis of post-stroke shoulder-hand syndrome

Exclusion criteria:

* Acute bursitis, tendonitis or tendon tear
* Fracture, dislocation or joint infection within 3 months
* Malignancy at treatment site
* Seizure
* Prosthesis or implant at treatment site
* Pregnancy

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
pain | 0,7, 14,28 days
  change of 10-point Visual Analog Scale (0-10, higher scores mean a worse outcome)

SECONDARY OUTCOMES:
strength of upper limb | 0,7, 14,28 days
  change of score of Manual muscle testing (0-5, higher scores mean a better outcome)
spasticity of upper limb | 0,7, 14,28 days
  change of Modified Ashworth Scale (0-4, higher scores mean a worse outcome)
range of motion of shoulder | 0,7, 14,28 days
  Change in range of motion in degree in flexion, extension, abduction, external and internal rotation (0-180 degrees,higher scores mean a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Ming Yen Y Hsiao, MDPHD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan